CLINICAL TRIAL: NCT04397835
Title: Psychological Impact of Quarantine During the COVID-19 Outbreak and Worsening of Cardiovascular Risk in the French General Population: a Prospective Cohort Study
Brief Title: Psychological Impact of COVID-19 Quarantine and Worsening of Cardiovascular Risk in the French General Population
Acronym: PSYCOV-CV
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0135
Record Dates: First submitted 2020-04-21; First posted 2020-05-21 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: COVID-19; Anxiety; Depression; Stress
Keywords: quarantine; psychological impact; cardiovascular disease; general population
MeSH Terms: conditions — COVID-19; Anxiety Disorders; Depression; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In response to the COVID-19 outbreak, the French government put in place home quarantine of the general population in order to limit the transmission of the virus. It is obvious that quarantine at home have a psychological impact which could worsened cardiovascular risk. Our aim is to assess risk factors for severe stress, anxiety or depression, during and after quarantine, as well as risk factors (including stress, anxiety or depression), in the worsening of cardiovascular risk.

DETAILED DESCRIPTION:
In response to the COVID-19 outbreak, the French government put in place home quarantine of the general population in order to limit the transmission of the virus. It is obvious that quarantine at home have a psychological impact which could worsened cardiovascular risk. Our aim is to assess risk factors for severe stress, anxiety or depression, during and after quarantine, as well as risk factors (including stress, anxiety or depression), in the worsening of cardiovascular risk.

A prospective epidemiological observational cohort study will be carried out (in French general population aged 50 to 89 years) with data collection by telephone interviews (in agreement with the context of quarantine).

The telephone interviews will be carried out during quarantine (V1), in the month following the end of quarantine (V2) and then, at 6 (V3) and 12 (V4) months. At baseline, the questionnaire will focus on socio-demographic and contextual characteristics related to the COVID-19 outbreak, medical history, cardiovascular risk factors and treatments, anxiety and depression scales. Next (after the quarantine), the questionnaire will focus on the evolution of cardiovascular risk factors and the occurrence of acute cardiovascular events, the evolution of treatments and post-traumatic stress, anxiety or depression scales.

The assessment of risk factors for severe stress, anxiety or depression, during and after quarantine, as well as risk factors of the worsening of cardiovascular risk will be based on mixed logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* All participants of the MONALISA survey residing in south-western France (Toulouse area).

Exclusion Criteria:

* Opposition to participate in this new survey
* Pregnancy or breastfeeding
* Subject under guardianship, curatorship or safeguard of justice
* Lack of health insurance coverage

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A sample of 1600 subjects was randomly recruited from the general population to participate in the MONALISA cross-sectional surveys on the prevalence of cardiovascular risk factors in 2005. Men and women aged 35-74, living in Toulouse area, were recruited between 2005 and 2008.
  The participants of the MONALISA population survey had agreed to be contacted, after the end of the MONALISA study, to take news of their state of health.
  Considering that the participation rate of the people contacted will be high (greater than 70%, taking into account the quarantine context), more than 800 participants (now aged 50 to 89 years) should be able to be included.
Sampling Method: Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-07-17 (Actual)

PRIMARY OUTCOMES:
worsening of cardiovascular risk (treatments) | at 1, 6 and 12 month
  The worsening of the cardiovascular risk factors during or after quarantine (versus before quarantine) will be considered in case of:
  - introduction or increase of antihypertensive, lipid-lowering or hypoglycaemic drug treatment on the prescription
worsening of cardiovascular risk (smoking consumption) | at 1, 6 and 12 month
  The worsening of the cardiovascular risk factors during or after quarantine (versus before quarantine) will be considered in case of increased smoking consumption
worsening of cardiovascular risk (food balance) | at 1, 6 and 12 month
  The worsening of the cardiovascular risk factors during or after quarantine (versus before quarantine) will be considered in case of alteration of the food balance
worsening of cardiovascular risk (weight gain) | at 1, 6 and 12 month
  The worsening of the cardiovascular risk factors during or after quarantine (versus before quarantine) will be considered in case of weight gain
worsening of cardiovascular risk (physical activity) | at 1, 6 and 12 month
  The worsening of the cardiovascular risk factors during or after quarantine (versus before quarantine) will be considered in case of:
  - reduction in the level of physical activity

SECONDARY OUTCOMES:
psychological impact of the quarantine on anxiety | at 1, 6 and 12 month
  " Generalized Anxiety Disorder " (GAD-7) : Spitzer, R. L., Kroenke, K., Williams, J. B. W. et Löwe, B. (2006). A brief measure for assessing generalized anxiety disorder: The GAD-7. Archives of Internal Medicine, 166(10), 1092-1097.
psychological impact of the quarantine on health | at 1, 6 and 12 month
  "Patient Health Questionnaire " (PHQ-9) : Kroenke, K., Spitzer, R. L. et Williams, J. B. W. (2001). The PHQ-9: Validity of a brief depression severity measure. J Gen Intern Med, 16(9), 606-613.
psychological impact of the quarantine on stress | at 1, 6 and 12 month
  " Impact of Event Scale - Revised " (IES-R) :
  * Weiss, D. S. et Marmar, C. R. (1996). The Impact of Event Scale-Revised. Dans J. P. Wilson et T. M. Keane (dir.). Assessing psychological trauma and PTSD. New York : Guildford Press.
  * Brunet, A., St-Hilaire, A., Jehel, L. et King, S. (2003). Validation of a French Version of the Impact of Event Scale-Revised.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Bérard, Principal Investigator — Service d'Epidémiologie, CHU de Toulouse UMR 1027, INSERM
Locations (1):
- CHU de Toulouse, Toulouse, Occitanie, France